CLINICAL TRIAL: NCT02152527
Title: Myocardial Energetics as a Target for Treatment of Ischemic Heart Disease: A Translational Approach From Patient to Mitochondria
Brief Title: Prospective Observational Study of Trimetazidine Influence on Mitochondrial Metabolism in Human Heart Ventricle
Status: Completed | Type: Observational
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Marko Ljubkovic, associate professor, M.D., PhD, University of Split, School of Medicine
Other Study IDs: TMZHHV
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Parts of human left ventricular muscle
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trimetazidine: Patients for coronary artery bypass grafting surgery who had preoperative trimetazidine usage in standard ischemic coronary disease therapy.
- Control: Patients for coronary artery bypass grafting surgery who had standard therapy for ischemic coronary disease without trimetazidine.

SUMMARY:
Trimetazidine (1-[2,3,4-trimethoxybenzyl] piperazine dihydrochloride) is a clinically effective antianginal agent. Despite these clinical successes, the understanding of trimetazidine's mechanism of action remains incomplete, particularly influence of trimetazidine on mitochondrial function in isolated human cardiomyocytes. The investigators will perform this study to seek possible differences in mitochondrial respiration related to standard preoperative enrolled trimetazidine therapy.

DETAILED DESCRIPTION:
Background:

Different types of medication are used for treatment of ischemic heart disease. One of recently developed drugs is trimetazidine. Although it clinical benefits are clear, mechanism by which this occurs is as yet undefined. In few animal studies authors try to define what effects trimetazidine has on both fatty acid and glucose metabolism in heart. Data collected from human cardiomyocytes are rare. Available data suggest that trimetazidine may act as a potent inhibitor of beta oxidation, with no significant effect on glucose oxidation.

Objective:

Primary objective: collection of mitochondrial respiration data using human heart ventricular samples. Secondary objective: define possible differences in mitochondrial respiration depending on preoperative trimetazidine usage.

Methods:

Regularly scheduled patients for coronary artery bypass grafting surgery who accept to participate in study will be enrolled in further protocol. Patients with inclusion criteria and without exclusion criteria will be enrolled in the study. At the end of operation, surgeon will take biopsy sample of left ventricle for mitochondrial function and metabolic activity analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease who are candidates for coronary artery bypass graft (CABG) surgery.

Exclusion Criteria:

* Emergency patients, patients who already had heart surgery, patients with acute coronary syndrome in last 2 months, patients with inability to understand patient information and informed consent.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease planned for coronary artery bypass grafting
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in rate of myocardial oxygen consumption expressed in pmolO2/min/units of citrate synthase activity. | Within 24 hours after tissue biopsy
  Investigators will obtain left ventricular biopsy samples from patients suffering from ischemic heart disease. Samples will be prepared in the laboratory for the purpose of assessment of mitochondrial respiration. Using the specific substrates from either fatty acid or carbohydrate metabolic pathways will enable investigation of the effect of trimetazidine on cardiac tissue metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Ljubković, M.D., PhD, Principal Investigator — Department of Physiology, University of Split School of Medicine
Locations (1):
- School of Medicine, University of Split, Split, Croatia